CLINICAL TRIAL: NCT04795843
Title: MovetheHip-trial: The Effectiveness of Exercise and Patient Education Compared With Usual Care on Self-reported Pain in Patients With Hip Dysplasia
Brief Title: Exercise and Patient Education Compared With Usual Care in Patients With Hip Dysplasia
Acronym: MovetheHip
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Research Unit for General Practice, Aarhus University (Other); VIA University College (Other); Copenhagen University Hospital, Hvidovre (Other); Defactum, Central Denmark Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MovetheHip
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Hip Dysplasia
Keywords: Hip Dislocation, Congenital; Exercise; Patient education; Usual care; Effectiveness; Cost-effectiveness; Process evaluation; Periacetabular osteotomy
MeSH Terms: conditions — Hip Dislocation; Hip Dislocation, Congenital; Motor Activity | interventions — Exercise; Patient Education as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise and patient education (Experimental): 6-months
  Interventions: Other: Exercise and patient education
- Usual Care (Active Comparator): 6-months
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Exercise and patient education — Over a period of 6-months, patients will be offered eight one-to-one supervised training sessions. In these sessions, patients will be instructed in a home-based exercise programme and given patient education. The programme includes four exercises covering strength and stability training. The exercises will be performed in sets of three with a minimum of 5 repetitions, and patients will be instructed to perform a minimum of three training sessions each week. Each of the exercises can be progressed through three levels of difficulty, allowing for individualised treatment with regard to exercise quality and perceived exertion according to the Borg CR10 scale. Exercises will be performed on a perceived exertion level from somewhat hard (level 5) to very hard (level 7). Patient education includes pain management, a focus on exercise adherence and progression, and advice on physical activity.
  Arms: Exercise and patient education
Other: Usual Care — Patients will follow usual care, including an individual consultation on self-management of hip symptoms and general advice on exercise and physical activity.
  Arms: Usual Care

SUMMARY:
This effectiveness trial will investigate if patients with hip dysplasia randomised to exercise and patient education have a different mean change in self-reported pain measured by the Copenhagen Hip and Groin Outcome Score (HAGOS) compared with those randomised to usual care over a six-month follow-up period.

Participating patients will be allocated to either exercise and patient education or usual care. Alongside this, a health-economic study and a process-evaluation study will be conducted.

DETAILED DESCRIPTION:
This study is a parallel-group superiority randomised controlled trial. Alongside this, a health-economic study and a process-evaluation study will be conducted. Participating patients will be allocated to either exercise and patient education or usual care at a 1:1 ratio. The primary outcome is change in self-reported pain measured with Copenhagen Hip and Groin Outcome Score (HAGOS) from baseline to 6-month follow-up.

The effectiveness of exercise and patient education compared with usual care will be reported in the primary trial paper, including the primary outcome and the following secondary outcomes: HAGOS symptoms, HAGOS function in daily living (ADL), HAGOS function in sport and recreation (sport/recreation), HAGOS participation in physical activity (participation), HAGOS quality of life (QOL), the impact of hip disease with the Short Version of the International Hip Outcome Tool (iHOT-12), lower limb reach length (anterior, posteromedial, posterolateral), single-leg hip for distance (SLHD) test and hip muscle strength (flexion, extension and abduction).

The primary aim of this effectiveness trial is to investigate if patients with hip dysplasia randomised to exercise and patient education have a different mean change in self-reported pain measured by the Copenhagen Hip and Groin Outcome Score (HAGOS) compared with those randomised to usual care over a six-month follow-up period.

The primary hypothesis: Patients randomised to exercise and patient education will have a between-group mean change score on the HAGOS pain that is at least 10 points higher than those randomised to usual care over a 6-month follow-up period.

The secondary aims are to compare mean changes between the two groups on the other HAGOS subscales over a 6-month follow-up period. Similar comparisons will be made on self-reported mean changes in the Short Version of the International Hip Outcome Tool (iHOT-12) and mean changes in performance, balance and hip muscle strength.

A full trial protocol will be published and made publicly available. All primary and secondary outcomes will be analysed with the intention-to-treat principle. Between-group differences from baseline to 3-month and 6-month follow-up of continuous outcomes will be estimated using repeated measurement analysis in a mixed-effects model, including patient as a random effect, with a fixed factor for group and time and the corresponding interaction (Group × Time), adjusted for baseline values. Between-group differences of continuous outcomes from baseline to 6-month follow-up will be analysed with an unpaired t-test, where between-group differences of categorical data from baseline to 6-month follow-up will be analysed with a binominal regression model using risk difference as a measure of association. In this paper, all collected outcomes will be listed, and it will be described that the below listed will be reported in other papers (i.e. health-economic study and process-evaluation study) and secondary papers.

In the health-economic study, the investigators will investigate the cost-utility and cost-effectiveness of exercise and patient education compared with usual care over 12 months. Outcomes for this paper will be measured at baseline, 3-, 6-, 9- and 12-month follow-up. Incremental cost-effectiveness ratios (ICER) will be calculated by dividing the difference in costs by the difference in effects (quality-adjusted life years and HAGOS pain). The uncertainty around the ICER and 95% confidence intervals (CIs) surrounding the cost differences will be estimated with 95% bootstrapped CIs based on non-parametric bootstrapping and will be graphically presented on cost-effectiveness planes and cost-effectiveness acceptability curves.

In the process-evaluation study, the investigators will explore the functioning of the intervention by evaluating the implementation, mechanisms of change and the contribution of contextual factors over 6 months.

Implementation includes the implementation process, fidelity, dose and reach. The implementation process will evaluate the structures and resources through which delivery is achieved. Fidelity aspects will evaluate the extent to deliver each component as planned and registered during the intervention period using self-report questionnaires. The dose will evaluate how much intervention is delivered and registered during the intervention period using routine monitoring forms, and reach will be evaluated as patterns in uptake and adherence by baseline patient characteristics registered before and during the intervention period. Mechanisms of change include interactions between the intervention, the intervention providers and the patients. Interactions will be evaluated through four semi-structured focus group interviews with the intervention providers and the expert team (study coordinator, Kristian Thorborg and Julie S. Jacobsen) and quantitative data on reasons for not receiving surgery. Contextual factors will include events, personal understandings and interactions and their possible influence on the implementation. Contextual factors will be evaluated through one-to-one semi-structured interviews during and after the intervention period with 15-20 patients in the intervention group. Findings from quantitative and quantitative analyses will be merged, interpreted and reported jointly.

The below listed will be reported in secondary papers with a clear reference to the primary trial paper and trial registration, and it will hold "secondary analyses from a randomised controlled trial" in the title.

By using subgroup stratification, we will explore if muscle-tendon pain and pain sensitisation modify between-group changes of the primary and secondary outcomes over 6 months. Furthermore, we plan to conduct an instrumental variable analysis on primary and secondary outcomes in an attempt to investigate the efficacy of the intervention. These analyses will be reported in secondary papers with clear reference to the primary trial paper.

In addition, the investigators plan to evaluate the psychometric properties of HAGOS and iHOT-12 in patients with hip dysplasia, and finally, the investigators plan to describe if hip osteoarthritis progresses over 5 and 10 years using the Tönnis osteoarthritis classification.

ELIGIBILITY:
Inclusion Criteria:

* Radiographically verified hip dysplasia by a Wiberg's centre edge (CE) angle of 10-25 degrees and an acetabular Index (AI) angle >10 degrees
* Hip and/or groin pain as primary pain for at least three months
* Candidate for periacetabular osteotomy (PAO) but unwilling to undergo PAO, or on a waiting list for surgery (PAO) for 12 months or longer
* Not candidate for PAO (negative impingement test, BMI >25, hip osteoarthritis, age >45 years or reduced hip range of motion)

Exclusion Criteria:

* Self-reported pain score >80 points measured with Copenhagen Hip and Groin outcome score
* Any major planned surgery (i.e. arthroplastic surgery or discectomy surgery)
* BMI >35
* Acetabular retroversion defined by crossover sign and posterior wall sign
* Calvé Legg Perthes or epiphysiolysis
* Previous pelvic/hip surgery in index limb
* Previous pelvic/hip surgery within the last 2 years in contralateral limb
* Previous surgery due to herniated disc or spondylodesis
* Previous arthroplastic surgery in the hip, knee or ankle
* Physical (pregnancy/trauma), neurological, medical or rheumatic conditions severely affecting the hip function
* Inadequacy in written and spoken Danish, mental illness or other conditions affecting the ability to follow mandatory procedures for participation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-04-16 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in self-reported pain measured with The Copenhagen Hip and Groin Outcome Score (HAGOS) (continuous data) | From baseline to 6-month follow-up. Outcome measured at baseline, 3- and 6-month follow-up. In addition at 9- and 12-month follow-up (health economic study) and after 2, 5 and 10 years (describing if hip osteoarthritis progresses over time)
  HAGOS pain sub-item measures degree of hip and/or groin pain through ten individual questions on a score from 0 to 100, higher score indicates lower pain.

SECONDARY OUTCOMES:
Change in self-reported symptoms measured with HAGOS (continuous data) | From baseline to 6-month follow-up. Outcome measured at baseline, 3- and 6-month follow-up. In addition at 9- and 12-month follow-up and after 2, 5 and 10 years (describing if hip osteoarthritis progresses over time)
  HAGOS symptoms sub-item measures hip and/or groin symptoms and difficulties through seven individual questions on a score from 0 to 100, higher score indicates lower symptoms.
Change in self-reported physical function, daily living (ADL) measured with HAGOS (continuous data) | From baseline to 6-month follow-up. Outcome measured at baseline, 3- and 6-month follow-up. In addition at 9- and 12-month follow-up and after 2, 5 and 10 years (describing if hip osteoarthritis progresses over time)
  HAGOS ADL sub-item measures degree of difficulty due to hip and/or groin problems through five individual questions on a score from 0 to 100, higher score indicates higher function.
Change in self-reported physical function in sports and recreational activities (sport/recreation) measured with HAGOS (continuous data) | From baseline to 6-month follow-up. Outcome measured at baseline, 3- and 6-month follow-up. In addition at 9- and 12-month follow-up and after 2, 5 and 10 years (describing if hip osteoarthritis progresses over time)
  HAGOS sport/recreation sub-item measures degree of difficulty due to hip and/or groin problems through eight individual questions on a score from 0 to 100, higher score indicates higher function.
Change in self-reported participation in physical activities (participation) measured with HAGOS (continuous data) | From baseline to 6-month follow-up. Outcome measured at baseline, 3- and 6-month follow-up. In addition at 9- and 12-month follow-up and after 2, 5 and 10 years (describing if hip osteoarthritis progresses over time)
  HAGOS participation sub-item measures how degree of ability to participate in physical activities is affected by hip and/or groin problems through two individual questions on a score from 0 to 100, higher score indicates higher ability to participate in physical activities.
Change in self-reported quality of life (QOL) measured with HAGOS (continuous data) | From baseline to 6-month follow-up. Outcome measured at baseline, 3- and 6-month follow-up. In addition at 9- and 12-month follow-up and after 2, 5 and 10 years (describing if hip osteoarthritis progresses over time)
  HAGOS QOL sub-item measures hip-related quality of life through five individual questions on a score from 0 to 100, higher score indicates higher quality of life.
Change in impact of hip disease using the Short Version of the International Hip Outcome Tool (iHOT- 12) (continuous data) | From baseline to 6-month follow-up. Outcome measured at baseline and 6-month follow-up. In addition at 12-month follow-up and after 2, 5 and 10 years (describing if hip osteoarthritis progresses over time)
  iHOT-12 measures impact of hip disease in young, active patients through 12 questions on a score from 0-100.
Change in anterior lower limb reach distance measured with the Y-balance test (continuous data) | From baseline to 6-month follow-up. Outcome measured at baseline and 6-month follow-up
  Anterior lower limb reach distance measures functional performance when maintaining balance on one leg, reported in cm normalised to limb length.
Change in posteromedial lower limb reach distance measured with the Y-balance test (continuous data) | From baseline to 6-month follow-up. Outcome measured at baseline and 6-month follow-up
  Posteromedial lower limb reach distance measures functional performance when maintaining balance on one leg, reported in cm normalised to limb length.
Change in posterolateral lower limb reach distance measured with the Y-balance test (continuous data) | From baseline to 6-month follow-up. Outcome measured at baseline and 6-month follow-up
  Posterolateral lower limb reach distance measures functional performance when maintaining balance on one leg, reported in cm normalised to limb length.
Change in single-leg jump distance measured with single-leg hop for distance test (continuous data) | From baseline to 6-month follow-up. Outcome measured at baseline and 6-month follow-up
  Single-leg jump test measures functional performance when jumping on one leg, reported in cm normalised to height.
Change in isometric hip flexion strength using a dynamometer with external belt-fixation (continuous data) | From baseline to 6-month follow-up. Outcome measured at baseline and 6-month follow-up
  Isometric hip flexion test measures isometric maximum voluntary contraction (MVC) in sitting position. Strength values will be normalised to moment arms and weight and reported in Nm/kg bodyweight.
Change in isometric hip extension strength using a dynamometer with external belt-fixation (continuous data) | From baseline to 6-month follow-up. Outcome measured at baseline and 6-month follow-up
  Isometric hip extension test measures isometric maximum voluntary contraction (MVC) in prone position. Strength values will be normalised to moment arms and weight and reported in Nm/kg bodyweight.
Change in isometric hip abduction strength using a dynamometer with external belt-fixation (continuous data) | From baseline to 6-month follow-up. Outcome measured at baseline and 6-month follow-up
  Isometric hip abduction test measures isometric maximum voluntary contraction (MVC) in supine position. Strength values will be normalised to moment arms and weight and reported in Nm/kg bodyweight.

OTHER OUTCOMES:
Self-reported acceptable symptom state using the Patient Acceptable Symptom State (PASS) (dichotome data) | Measured at 6- and 12-month follow-up
  PASS measures perceived state of current hip and/or groin symptoms by the following question: Taking into account all the activities the patients are doing in their daily life, their level of pain, and also their functional impairments, do the patients consider that their current state of symptoms is acceptable (yes/no)?
Change in self-reported hip and/or groin pain intensity measured with a 100 mm Visual Analogue Scale (VAS) for pain in rest (continuous data) | From baseline to 6-month follow-up. Outcome measured at baseline, 6- and 12-month follow-up
  Hip and/or groin pain is measured on an electronic VAS from 0 to 100 mm within the last week.
Change in self-reported hip and/or groin pain intensity measured with a 100 mm Visual Analogue Scale (VAS) for pain during physical activity (continuous data) | From baseline to 6-month follow-up. Outcome measured at baseline, 6- and 12-month follow-up
  Hip and/or groin pain is measured on an electronic VAS from 0 to 100 mm within the last week.
Change in self-reported back pain intensity measured with a 100 mm Visual Analogue Scale (VAS) for pain in rest (continuous data) | From baseline to 6-month follow-up. Outcome measured at baseline, 6- and 12-month follow-up
  Back pain is measured on an electronic VAS from 0 to 100 mm within the last week.
Change in self-reported back pain intensity measured with a 100 mm Visual Analogue Scale (VAS) for pain in activity (continuous data) | From baseline to 6-month follow-up. Outcome measured at baseline, 6- and 12-month follow-up
  Back pain is measured on an electronic VAS from 0 to 100 mm within the last week.
Trust in the capability of the hip with a 100 mm Visual Analog Scale (0-100, 100 best) for trust during the single-leg hop for distance test (continuous data) | From baseline to 6-month follow-up. Outcome measured at baseline and 6-month follow-up
  Trust in the capability is measured immediately after the single-leg hop for distance test
Change in self-reported hip and/or groin pain during hip flexion strength test measured on a numerical rating scale (NRS) for pain (categorical data) | From baseline to 6-month follow-up. Outcome measured at baseline and 6-month follow-up
  Hip and/or groin is measured immediately after isometric hip flexion strength test
Change in self-reported hip and/or groin pain during hip extension strength test measured on a numerical rating scale (NRS) for pain (categorical data) | From baseline to 6-month follow-up. Outcome measured at baseline and 6-month follow-up
  Hip and/or groin is measured immediately after isometric hip extension strength test
Change in self-reported hip and/or groin pain during hip abduction strength test measured on a numerical rating scale (NRS) for pain (categorical data) | From baseline to 6-month follow-up. Outcome measured at baseline and 6-month follow-up
  Hip and/or groin is measured immediately after isometric hip abduction strength test
Change in self-reported usage of analgesics (y/n/type/dose) | From baseline to 6-month follow-up. Outcome measured at baseline and 6-month follow-up
  Analgesics include paracetamol/acetaminophen, ibuprofen and other NSAIDs, and morphine/opioids.
Number of serious adverse events (SAE) and adverse events (AE) related to the interventions, clinical assessments or conduct of the trial within the intervention period (continuous data) | From baseline to 6-month follow-up.
  SAE and AE that may occur within the intervention period will be identified in different ways: by self-reporting by the patients and by observation from the intervention providers and test physiotherapists. Furthermore, a short patient-reported questionnaire at the 3- and 6- month follow-up will be used to ensure that all SAE and AE requiring medical treatment will be recorded. In addition, the included patients will be encouraged to report health issues and injuries affecting adherence to allocated treatments to the principal investigator within the intervention period.
Adherence measured by the 6-item Exercise Adherence Rating Scale (EARS) (continuous data) | From baseline to 6-month follow-up. Outcome measured at 3- and 6-month follow-up
  Adherence is scored on a scale from 0 to 24 points by the patients, 24 indicating full adherence
Adherence measured at number of completed training sessions (continuous data) | From baseline to 6-month follow-up. Outcome measured every week.
  Number of completed training sessions is reported prospectively by the patients in standardised registration forms (range 0-78)
Change in quality-adjusted life years (QALYs) measured with EuroQoL 5-dimension (EQ-5D-5L) and valued using preference weights (continuous data) | From baseline to 12-month follow-up. Outcome measured at baseline, 3-, 6-, 9- and 12-month follow-up
  The EQ-5D-5L is a five-item patient-reported outcome measure designed to assess generic health-related quality-of-life. We will used the UK value set in this study, because a Danish value set is not yet available. These values range from -0.285 to 1.0, a value of 1.0 corresponds to full health, 0 corresponds to death and negative values correspond to health status considered to be worse than death. QALYs will be reported in the health economic study.
Productivity loss measured with Productivity Costs Questionnaire (IPCQ) (continuous data) | From baseline to 6-month follow-up. Outcome measured at baseline, 3-, 6-, 9- and 12-month follow-up
  The IPCQ questionnaire includes three modules measuring productivity losses of paid work due to 1) absenteeism and 2) presenteeism and productivity losses related to 3) unpaid work. Productivity loss will be reported in the health economic study.
Change in muscle-tendon pain in the iliopsoas measured with a pain-provocation test (dichotomous data) | From baseline to 6-month follow-up. Outcome measured at baseline and 6-month follow-up
  The iliopsoas pain-provocation test measured known pain palpatory pain in the muscle through the lower lateral part of the abdomen and/or just distal to the inguinal ligament. Muscle-tendon pain will be reported in a secondary paper.
Change in muscle-tendon pain in the abductors measured with a pain-provocation test (dichotomous data) | From baseline to 6-month follow-up. Outcome measured at baseline and 6-month follow-up
  The abductor pain-provocation test measured known palpatory pain at the insertion point at the greater trochanter and pain with side-lying abduction against resistance. Muscle-tendon pain will be reported in a secondary paper.
Change in temporal summation of pain (TS) at the hip (continuous data) | From baseline to 6-month follow-up. Outcome measured at baseline and 6-month follow-up
  TS measures increase in pain recorded on a numerical rating scale (NRS) (range 0-10) as the difference in pain rating between a single pinprick stimuli and a train of 10 pinprick stimuli applied to the rectus femoris muscle. TS will be reported in a secondary paper.
Change in temporal summation of pain (TS) at the forearm (continuous data) | From baseline to 6-month follow-up. Outcome measured at baseline and 6-month follow-up
  TS measures increase in pain recorded on a numerical rating scale (NRS) (range 0-10) as the difference in pain rating between a single pinprick stimuli and a train of 10 pinprick stimuli applied to the forearm. TS will be reported in a secondary paper.
Change in pressure pain threshold (PPT) at the hip (continuous data) | From baseline to 6-month follow-up. Outcome measured at baseline and 6-month follow-up
  PPT measures first sensation of pain when increasing pressure is applied with an algometer at the rectus femoris muscle, reported as kPa. PPT will be reported in a secondary paper.
Change in pressure pain threshold (PPT) at the forearm (continuous data) | From baseline to 6-month follow-up. Outcome measured at baseline and 6-month follow-up
  PPT measures first sensation of pain when increasing pressure is applied with an algometer at the forearm, reported as kPa. PPT will be reported in a secondary paper.
Change in osteoarthritis grade measured by the Tönnis osteoarthritis classification (categorical data) | From baseline to 5- and 10-years follow-up. Outcome measured at baseline and after 2, 5 and 10 years (describing if hip osteoarthritis progresses over time)
  Tönnis osteoarthritis classification grade degree of osteoarthritis from 0-3, and 0 indicates no signs of osteoarthritis and 3 indicates severe osteoarthritis described by large cysts, severe narrowing of the joint space, severe femoral head deformity, and avascular necrosis
Number of other treatments received by the patients (number and text) | From baseline to 12-month follow-up (Health economic study). Outcome measured at 3- 6-, 9- and 12-month follow-up and after 2, 5 and 10 years (describing if hip osteoarthritis progresses over time)
  Self-reported and registry-based data

CONTACTS AND LOCATIONS:
Overall Officials: Julie S Jacobsen, PhD, Principal Investigator — VIA University College; Inger Mechlenburg, DMSc, Study Director — Aarhus University Hospital; Kristian Thorborg, PhD, Study Chair — Copenhagen University Hospital, Hvidovre; Rasmus Ø Nielsen, PhD, Study Chair — University of Aarhus; Stig S Jakobsen, PhD, Study Chair — Aarhus University Hospital; Lisa G Oestergaard, PhD, Study Chair — Defactum, Central Denmark Region; Kjeld Søballe, PhD, Study Chair — Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Aarhus N
  - Silkeborg Regional Hospital., Silkeborg

IPD SHARING:
Plan to Share IPD: Yes
What data will be shared: All quantitative individual participant data collected during the trial, after deidentification.
  With whom will data be shared: Researchers who provide a methodologically sound proposal.
  For what types of analyses: To achieve aims in the approved proposal.
  The abovementioned is based on Data Sharing Statements for Clinical Trials: A Requirement of the ICMJE located at: http://www.icmje.org/news-and-editorials/data_sharing_june_2017.pdf.
Supporting Information: Study Protocol, SAP
Time Frame: Immediately following publication and ending 5 years following primary article publication.
Access Criteria: Proposals should be directed to jsaj@via.dk. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Jacobsen JS, Evans R, Morgan K, Thorborg K, Oestergaard LG, Sorensen D. An exercise and patient education intervention to reduce pain and physical limitations in adults with acetabular dysplasia: study protocol for a process evaluation integrated within a randomised controlled trial (the MovetheHip trial). Trials. 2024 Jun 24;25(1):411. doi: 10.1186/s13063-024-08262-y. PMID 38915128
- [Background] Jacobsen JS, Thorborg K, Nielsen RO, Jakobsen SS, Foldager C, Sorensen D, Oestergaard LG, van Tulder MW, Mechlenburg I. Comparing exercise and patient education with usual care in the treatment of hip dysplasia: a protocol for a randomised controlled trial with 6-month follow-up (MovetheHip trial). BMJ Open. 2022 Sep 20;12(9):e064242. doi: 10.1136/bmjopen-2022-064242. PMID 36127096
- [Background] Jacobsen JS, Thorborg K, Sorensen D, Jakobsen SS, Nielsen RO, Oestergaard LG, Soballe K, Mechlenburg I. Feasibility and acceptability of a six-month exercise and patient education intervention for patients with hip dysplasia: A mixed methods study. Musculoskelet Sci Pract. 2022 Oct;61:102615. doi: 10.1016/j.msksp.2022.102615. Epub 2022 Jun 24. PMID 35820302